CLINICAL TRIAL: NCT03959124
Title: The Effect of Deep Brain Stimulation on Memory Network and Neurological Function of Alzheimer's Disease
Brief Title: Deep Brain Stimulation for Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Collaborators: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB106-68-A
Record Dates: First submitted 2019-02-21; First posted 2019-05-22 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-06

CONDITIONS: Alzheimer Disease; Dementia, Alzheimer Type; Deep Brain Stimulation
Keywords: magnetic resonance image
MeSH Terms: conditions — Alzheimer Disease | interventions — Deep Brain Stimulation; Amyloid beta-Protein Precursor; Rivastigmine; Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AD with DBS (Experimental): Alzheimer's disease subjects with optimal medication therapy and with DBS treatment
  Interventions: Device: Deep brain stimulation; Drug: Best medical treatment for Alzheimer's disease
- AD without DBS (Active Comparator): Alzheimer's disease subjects with optimal medication therapy and without DBS treatment
  Interventions: Drug: Best medical treatment for Alzheimer's disease
- Normal control (No Intervention): Matched aged and demographics subjects

INTERVENTIONS:
Device: Deep brain stimulation — Brain stimulation electrodes at parameters 2.0~4.5 V；60 μs；20 Hz
  Other Names: Deep brain stimulation electrodes (Medtronic or Abbott)
  Arms: AD with DBS
Drug: Best medical treatment for Alzheimer's disease — Alzheimer's disease patients take medications including Exelon (Rivastigmine Tartrate), Witgen (Memantine) for at least 3 months without plan of dosage adjustment
  Other Names: Exelon (Rivastigmine Tartrate), Witgen (Memantine)
  Arms: AD with DBS; AD without DBS

SUMMARY:
Background: Deep brain stimulation (DBS) is used to modulate the activity of dysfunctional brain circuits. The safety and preliminary efficacy of nucleus basalis of Meynert (NBM)-DBS in Alzheimer's disease (AD) is proved in a recent phase 1 clinical trial, yet, the mechanism still unknown.

Objective: 1. To compare the brain structure and functional circuits between a) AD patients with optimal drug treatment (ODT) plus NBM-DBS, b) AD with ODT and c) normal age-and sex-matched control. 2. To evaluate the clinical effectiveness of NBM-DBS in AD patients 60-75 year-old. 3. To evaluate the abnormal functional circuitry response to acute and chronic NBM-DBS in AD.

Methods: A total of 30 subjects (10 subjects of AD with ODT plus NBM-DBS; 10 subjects of AD with ODT and 10 subjects of normal age-and sex-matched subjects) will be enrolled in this prospective, with normal control, Phase II study. Study tools will include clinical rating batteries, structure and functional imaging of magnetic resonance (MR) and positron emission tomography (PET), and electroencephalogram (EEG).

Expected Results: NBM-DBS will be proved to be an safe and effective treatment modality in AD patients 60-75 year-old. Through multi-modal images and EEG analysis, the possible action mechanisms of NBM-DBS on memory circuit will be discussed. The study results may shed a light on this helpless neurodegenerative disease of dementia.

ELIGIBILITY:
Inclusion Criteria:

For groups (AD with/ without DBS)

1. Confirmed Alzheimer's dementia diagnosis
2. Regular medications taking for at least 3 months
3. Clinical Dementia Rating: 0.5 - 2
4. Mini Mental Status Examination: ≦ 26
5. Amyloid PET: positive
6. Informed consent signed by patients or families

For normal control group

1. No cognitive impairment (Mini Mental Status Examination)
2. Amyloid PET: negative
3. Informed consent signed by patients and families

Exclusion Criteria:

For groups (AD with/ without DBS)

1. Structural lesions identified by Magnetic resonance imaging (ex: stroke, brain surgery)
2. Other neurodegenerative/ neuropsychiatric diseases
3. Systemic medical diseases with cognitive impairment (ex: anemia, thyroid disease)
4. Can't have regular follow-up visit

For normal control group

1. Structural lesions identified by Magnetic resonance imaging (ex: stroke, brain surgery)
2. Dementia/ neurodegenerative/ neuropsychiatric diseases
3. Systemic medical diseases with cognitive impairment (ex: anemia, thyroid disease)
4. Can't have regular follow-up visit

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-04-06 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) | One year
  Change from baseline in Alzheimer's Disease Assessment Scale-cognitive subscale; Total scores range from 0-70. Higher scores (≥ 18) indicate worse cognitive function. It consists of 11 tasks measuring the disturbances of memory, language, praxis, attention and other cognitive abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Yuan Chen, MD., Principal Investigator — Buddhist Tzu Chi General Hospital
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuhn J, Hardenacke K, Lenartz D, Gruendler T, Ullsperger M, Bartsch C, Mai JK, Zilles K, Bauer A, Matusch A, Schulz RJ, Noreik M, Buhrle CP, Maintz D, Woopen C, Haussermann P, Hellmich M, Klosterkotter J, Wiltfang J, Maarouf M, Freund HJ, Sturm V. Deep brain stimulation of the nucleus basalis of Meynert in Alzheimer's dementia. Mol Psychiatry. 2015 Mar;20(3):353-60. doi: 10.1038/mp.2014.32. Epub 2014 May 6. PMID 24798585
- [Background] Gratwicke J, Zrinzo L, Kahan J, Peters A, Beigi M, Akram H, Hyam J, Oswal A, Day B, Mancini L, Thornton J, Yousry T, Limousin P, Hariz M, Jahanshahi M, Foltynie T. Bilateral Deep Brain Stimulation of the Nucleus Basalis of Meynert for Parkinson Disease Dementia: A Randomized Clinical Trial. JAMA Neurol. 2018 Feb 1;75(2):169-178. doi: 10.1001/jamaneurol.2017.3762. PMID 29255885
- [Background] Kumbhare D, Palys V, Toms J, Wickramasinghe CS, Amarasinghe K, Manic M, Hughes E, Holloway KL. Nucleus Basalis of Meynert Stimulation for Dementia: Theoretical and Technical Considerations. Front Neurosci. 2018 Sep 3;12:614. doi: 10.3389/fnins.2018.00614. eCollection 2018. PMID 30233297
- [Background] Kuhn J, Hardenacke K, Shubina E, Lenartz D, Visser-Vandewalle V, Zilles K, Sturm V, Freund HJ. Deep Brain Stimulation of the Nucleus Basalis of Meynert in Early Stage of Alzheimer's Dementia. Brain Stimul. 2015 Jul-Aug;8(4):838-9. doi: 10.1016/j.brs.2015.04.002. Epub 2015 Apr 18. No abstract available. PMID 25991080
- [Background] Canter RG, Penney J, Tsai LH. The road to restoring neural circuits for the treatment of Alzheimer's disease. Nature. 2016 Nov 10;539(7628):187-196. doi: 10.1038/nature20412. PMID 27830780
- [Background] Iaccarino HF, Singer AC, Martorell AJ, Rudenko A, Gao F, Gillingham TZ, Mathys H, Seo J, Kritskiy O, Abdurrob F, Adaikkan C, Canter RG, Rueda R, Brown EN, Boyden ES, Tsai LH. Gamma frequency entrainment attenuates amyloid load and modifies microglia. Nature. 2016 Dec 7;540(7632):230-235. doi: 10.1038/nature20587. PMID 27929004